CLINICAL TRIAL: NCT02713672
Title: Cost-effectiveness of CYP2D6 and CYP2C19 Genotyping in Psychiatric Patients in Curacao
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Centraal (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Parnassia (Unknown); Klinika Capriles (Unknown); Psychiaters Maatschap Antillen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 70-72600-98-005
Record Dates: First submitted 2016-02-23; First posted 2016-03-21 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: CYP2D6, Psychiatric Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Psychiatric patients with a CYP2D6 or CYP2C19 PM or IM genotype, using antidepressants or antipsychotics metabolized by CYP2D6 or CYP2C19
  Interventions: Other: Dose adjustment according to genotype
- Control group (No Intervention): Psychiatric patients with a CYP2D6 or CYP2C19 EM genotype using antidepressants or antipsychotics

INTERVENTIONS:
Other: Dose adjustment according to genotype — Patients in the intervention group received a dose adjustment according to their CYP2D6 or CYP2C19 genotype based on guidelines of the KNMP
  Arms: Intervention group

SUMMARY:
The cytochrome P450 (CYP) is a group of metabolic enzymes, from which the 2D6 and CYP2C19 polymorphisms are specifically related to the metabolism of psychiatric drugs. The prevalence of CYP2D6 and CYP2C19 polymorphisms differs among ethnicities. Depending on the number of functional alleles, individuals are classified as Poor Metabolizer (PM), Intermediate Metabolizer (IM), Extensive Metabolizer (EM) or Ultra Rapid Metabolizer (UM).

Research has suggested that PM genotype is a predisposing factor for antipsychotic-induced side-effects. Besides susceptibility for side effects and lower quality of life, also, a relationship between phenotype and costs of care has been shown.

Guidelines recommend that PM, IM and UM genotypes need dose adjustment, to optimize the effectiveness of the drug and/or to reduce side effects. No research has been done to investigate cost-effectiveness of implementation of genotyping in daily clinical psychiatric practice.

This study investigates the effectiveness of implementation of CYP2D6 and CYP2C19 genotyping in psychiatric patients in Curacao and analyzes the costs of genotyping versus health benefits.

DETAILED DESCRIPTION:
Subjects

This study is carried out on the Caribbean island Curacao and in the Netherlands. The population (approx. 150,000 inhabitants) of Curacao is mainly of Negroid descent. Participants were recruited from the Klinika Capriles, (the only psychiatric hospital on the island) the psychiatric ward in the prison (FOBA) and the psychiatric polyclinic on the island (Psychiaters Maatschap Antillen). The study protocol was approved by the Medical Ethical Review Board (Maastricht) and study participants gave written informed consent after explanation about the study.

Inclusion criteria were: (i) An Antillean ethnicity, defined in line with the Dutch Central Bureau of Statistics as birth on the former Dutch Antilles and birth of at least one parent on the former Dutch Antilles. (ii) Age 18 years or older. (iii) The use of an antipsychotic or antidepressant and (iv) informed consent.

All the patients were genotyped and grouped according to predicted phenotype for CYP2D6 and CYP2C19. Information about medication use was collected. Patients using CYP2D6 or CYP2C19 inhibiting medication according to Flockhart were selected. Enzyme activity scores of patients using a strong inhibitor were multiplied by 0 which meant they converted automatically to a PM phenotype. In patients using medium inhibitors, activity scores were multiplied by 0.5. This is a widely used and accepted method.

All prescribed antipsychotics were calculated to a "Defined Daily Dose" (DDD) as defined by the World Health Organization (WHO). For every patient the total equivalent of the DDD was calculated. In this way it was possible to analyse if there were differences in total dose of antipsychotics being used between the phenotype groups.

Patients who needed dose adjustment based on phenotype according to the Royal Dutch Association for the Advancement of Pharmacy were selected.

Patients who were selected were matched with controls on gender, age and depot or oral medication use. All participants received a 25 guilder gift token if they cooperated in the study at both measuring points.

Assessments

Subjective experience, psychopathology, extrapyramidal side effects, quality of life, global functioning and metabolic parameters were assessed at baseline (T0) and 4 months after dose adjustment (T1). A medical doctor, trainee in psychiatry, blind for the intervention, was responsible for all the measurements and was being trained in investigating extra pyramidal side effects and measuring global functioning. Patients receiving depot medication were measured in the same moment in the depot in T0 and T1.

Severity of patients' psychopathology was assessed with Brief Psychiatric Rating Scale (BPRS), which measures 24 symptoms of psychiatric disease and is validated in Dutch 20. Extrapyramidal symptoms were assessed with the St. Hans Ratings Scale (SHRS), which is a multidimensional rating scale for the evaluation of hyperkinesia, parkinsonism, akathisia and dystonia induced by neuroleptics. The dyskinesia is scored in two situations: in passive and active circumstances.

Akathisia was being measured by the Barnes Rating Scale (BARS) for Drug-Induced Akathisia. Subjective experience of the patients was measured with the Subjective Well-Being Under Neuroleptics Scale (SWN-20), which is a 20- item, self-rating scale which assesses the subjective experience over the preceding 7 days.

Quality of life was assessed with the EurolQol 5-D (EQ 5-D), which is a widely used rating scale, that measures health status on five dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression).

Global functioning was assessed with the World Health Organization Disability Assessment Schedule 2.0 (WHODAS-36) 36 item proxy-administered version. The questionnaire measures disability in 6 domains and was being administered by a personal care giver.

Metabolic parameters measured were blood pressure, Body Mass Index (BMI), waist size, cholesterol, High Density Lipo-protein (HDL), Low Density Lipo-protein (LDL), triglycerides, glucose, Hemoglobin A1c (HbA1C). Prolactin was also being measured. In patients receiving antipsychotics metabolized by CYP2D6, plasma levels of antipsychotics were measured.

Procedures

After baseline measurements, another medical doctor, trainee in psychiatry made dose adjustments according to guidelines of the Royal Dutch Association for the Advancement of Pharmacy (KNMP) which was updated July 2013. Generally three options were available: 1. Lowering/ enhancing the dose to 50-75% of the original dose 2. Prescription of medication not being metabolized by CYP2D6 or CYP2C19 3. Stop CYP2D6 or CYP2C19 inhibiting medication.

A standard procedure for dose adjustments was being followed: Lowering the dose was done in steps according to http://wiki.psychiatrienet.nl/index.php/SwitchAntipsychotics.

If an alternative antipsychotic had to be prescribed, first choice was flupentixol, second choice olanzapine, third choice quetiapine. Inhibiting medication meant to tranquilize was being replaced by benzodiazepines.

Complex cases were discussed with the research team and individual dose adjustment plans were being made.

ELIGIBILITY:
Inclusion Criteria:

1. Antillean ethnicity, defined in line with the Dutch Central Bureau of Statistics as birth on the former Dutch Antilles and birth of at least one parent on the former Dutch Antilles
2. age 18 years or older
3. use of an antipsychotic or antidepressant drug
4. written informed consent.

Exclusion Criteria:

1) no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
St Hans Rating Scale | 4 months
  Improvement on movement disorders
BPRS | 4 months
  Improvement on psychiatric symptoms
WHODAS 2.0 | 4 months
  Improvement on global functioning

SECONDARY OUTCOMES:
BMI | 4 months
  improvement in metabolic parameters
EQ 5D | 4 months
  Improvement in quality of life
SWN-20 | 4 months
  Improvement in subjective well-being under neuroleptics
blood pressure | 4 months
  Lowering of blood pressure
cholesterol spectrum | 4 months
  lowering of serum cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: Peter van Harten, Professor, Study Chair — GGZ Centraal; Wijbrand Hoek, Professor, Study Chair — Parnassia; David Vinkers, PhD, Study Chair — Maastricht University; Anne Koopmans, MD, Principal Investigator — Maastricht University
Locations (1):
- Zon en Schild, Amersfoort, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data about the individual CYP profiles is handed to involved clinicians after the research has finished

REFERENCES:
- [Derived] Koopmans AB, van Hoeken D, Clarke DE, Vinkers DJ, van Harten PN, Hoek HW. Proxy WHO Disability Assessment Schedule 2.0 Is Clinically Useful for Assessing Psychosocial Functioning in Severe Mental Illness. Front Psychiatry. 2020 Apr 15;11:303. doi: 10.3389/fpsyt.2020.00303. eCollection 2020. PMID 32351419
- [Derived] Koopmans AB, Vinkers DJ, Poulina IT, Gelan PJA, van Schaik RHN, Hoek HW, van Harten PN. No Effect of Dose Adjustment to the CYP2D6 Genotype in Patients With Severe Mental Illness. Front Psychiatry. 2018 Aug 7;9:349. doi: 10.3389/fpsyt.2018.00349. eCollection 2018. PMID 30131727